CLINICAL TRIAL: NCT06827665
Title: Clinical and Radiographic Evaluation of Allogenic Dentin Grafts for Alveolar Ridge Preservation: A Prospective Clinical Trial
Brief Title: Clinical and Radiographic Evaluation of Allogenic Dentin Grafts for Alveolar Ridge Preservation
Acronym: JUH
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jordan University Hospital (Other)
Collaborators: hanan Jafar (Unknown)
Responsible Party: Principal Investigator, Soukaina Ryalat, Principal Investigator, Jordan University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DDA-WTA-JUH
Record Dates: First submitted 2025-02-04; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Alveolar Ridge Preservation
MeSH Terms: interventions — bis(p-chlorophenyl)acetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DDA (Experimental): demineralized dentin allografts (DDA) will be given for alveolar ridge preservation, contributing to innovative, sustainable dental practices
  Interventions: Biological: DDA
- WTA (Experimental): Whole tooth allografts (WTA) will be given for alveolar ridge preservation, contributing to innovative, sustainable dental practices
  Interventions: Biological: WTA
- Control (No Intervention): Control

INTERVENTIONS:
Biological: DDA — : demineralized dentin allografts (DDA) allografts from human extracted teeth will be prepared and evaluated in a prospective clinical trial to assess their efficacy for alveolar ridge preservation. The reconstruction and preservation of the alveolar ridge after tooth extraction are essential for future prosthetic rehabilitation. Autogenous bone grafts, while effective, are limited by donor site morbidity and insufficient graft quantity. Allogenic dentin grafts, derived from healthy human donors, present a scalable solution.
  Other Names: demineralized dentin allografts (DDA)
  Arms: DDA
Biological: WTA — whole tooth allografts (WTA) allografts from human extracted teeth will be prepared and evaluated in a prospective clinical trial to assess their efficacy for alveolar ridge preservation. The reconstruction and preservation of the alveolar ridge after tooth extraction are essential for future prosthetic rehabilitation. Autogenous bone grafts, while effective, are limited by donor site morbidity and insufficient graft quantity. Allogenic dentin grafts, derived from healthy human donors, present a scalable solution.
  Other Names: Whole tooth allografts (WTA)
  Arms: WTA

SUMMARY:
For the first time, allografts from human-extracted teeth will be prepared and evaluated in a prospective clinical trial to assess their efficacy for alveolar ridge preservation. The reconstruction and preservation of the alveolar ridge after tooth extraction are essential for future prosthetic rehabilitation.

Autogenous bone grafts, while effective, are limited by donor site morbidity and insufficient graft quantity. Allogenic dentin grafts from healthy human donors present a scalable solution. This study aims to evaluate the biocompatibility and effectiveness of two types of allogenic dentin grafts-demineralized dentin allografts (DDA) and whole tooth allografts (WTA)-for alveolar ridge preservation, contributing to innovative, sustainable dental practices.

DETAILED DESCRIPTION:
This study holds significant importance for the fields of dentistry and maxillofacial surgery, addressing key clinical, scientific, and practical challenges:

1. Innovative Approach to Ridge Preservation o By evaluating allogenic dentin grafts for alveolar ridge preservation, this study introduces an innovative solution for post-extraction bone regeneration, offering a sustainable alternative to conventional grafting methods.
2. Addressing Limitations of Autogenous Grafts o Autogenous bone grafts, while effective, are limited by availability, patient acceptance, and donor site morbidity. Allogenic dentin grafts overcome these limitations, providing a readily available, safe, and effective option.
3. Sustainable Utilization of Extracted Teeth o Extracted teeth are typically discarded as biomedical waste. This study demonstrates their potential to be repurposed as valuable graft materials, promoting sustainability and reducing waste in dental practices.
4. Expanding the Body of Knowledge o There is limited research on allogenic dentin grafts compared to autogenous or xenogenic grafts. This study contributes valuable clinical and radiographic data, addressing a significant gap in the literature and paving the way for future research.
5. Clinical Relevance for Prosthetic Rehabilitation o Successful alveolar ridge preservation is critical for subsequent prosthetic treatments, including implants and dentures. This study provides evidence-based insights into new methods that improve outcomes for patients.
6. Potential for Broader Applications o By validating the efficacy of allogenic dentin grafts, this research supports the development of standardized protocols for their preparation and use, potentially expanding their application beyond ridge preservation to other bone regeneration procedures.
7. Encouraging Tissue Banking and Collaboration

ELIGIBILITY:
Inclusion and Exclusion Criteria for Donors:

Inclusion Criteria:

* Students, interns, or residents willing to participate and provide informed consent.
* No history of systemic diseases such as diabetes, hepatitis, or immune disorders.
* Negative blood screening for HIV, HBV, and HCV.
* Non-smokers or individuals who have not smoked within the last six months.

Exclusion Criteria:

* History of systemic conditions affecting oral or overall health.
* Positive blood tests for communicable diseases.
* Active oral infections or untreated dental caries.
* Pregnant or lactating individuals.
* Individuals with a history of smoking or substance abuse within the last six months.

Inclusion and Exclusion Criteria for Recipients:

Inclusion Criteria:

* Patients aged 18-60 years, requiring extraction of at least three teeth for clinical or therapeutic reasons.
* Patients in good systemic health without conditions that impair bone healing.
* Willingness to provide informed consent and participate in follow-ups.

Exclusion Criteria:

* Systemic conditions such as diabetes, osteoporosis, or immunodeficiency that could impair bone regeneration.
* Active oral infections at extraction sites.
* History of radiation therapy to the head and neck region.
* Smoking or smoking history within the last six months.
* Use of medications affecting bone metabolism (e.g., bisphosphonates, steroids).
* Pregnancy or lactation. Additional Justification for Extraction: Teeth chosen for extraction must meet one or more criteria:
* Severe periodontal disease.
* Irreversible pulpitis or structural damage.
* Non-restorable condition impacting oral health or functionality.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in alveolar ridge width and height (in mm) from baseline to 3 months post-extraction, measured using CBCT scans. | 3 months

SECONDARY OUTCOMES:
Change in alveolar crest height and width (in mm) from baseline to 3 months post-extraction, measured using CBCT scans, comparing DDA, WTA, and ungrafted control sites. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No